CLINICAL TRIAL: NCT07059481
Title: Evaluation of Oxidative Stress in Patients With Chronic Apical Periodontitis Treated With Single Session Root Canal Treatment Using Different Root Canal Sealers: in Vivo Study
Brief Title: Effect of Different Root Canal Sealers on Oxidative Stress Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: bengi gülgü (Other)
Responsible Party: Sponsor-Investigator, bengi gülgü, Principle Investigator, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/53
Record Dates: First submitted 2025-01-19; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Oxidative Stress; Chronic Apical Periodontitis
Keywords: oxidative stress; root canal sealers; chronic apical periodontitis; periapical index; total oxidant status; total antioxidant status; oxidative stress index; 8-epi; malondialdehyde; myeloperoxidase
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Intervention Model Description: the results obtained from the groups will be compared and correlated both within and between the groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: The root canal paste to be used will be selected from identical black envelopes by another physician who will not participate in the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- Bioceramic Group (Experimental): Patients which had been used bioceramic-based sealer (MTA Bioseal, Itena, France) while root canal treatment.
  Interventions: Other: Root Canal Treatment and Sample Collection; Diagnostic Test: PAI Score Comparasion
- 2- Epoxy amine Group (Experimental): Patients which had been used epoxyamine resin-based sealer (Itena Obturys, Itena, France) while root canal treatment.
  Interventions: Other: Root Canal Treatment and Sample Collection; Diagnostic Test: PAI Score Comparasion

INTERVENTIONS:
Other: Root Canal Treatment and Sample Collection — Single session root canal treatment procedure will be performed with VDW Gold Reciproc device and reciprocal files (Endo T-Must, Dentac, Turkey). Endodontium Samples will be collected from each patient's root canal, with 15 Hedström files (Dentsplay).
  Other Names: Saliva Sample Collection (two times per patient); Sample Collection from Endodontium while root canal treatment session.; Completion of root canal obturation with epoxyamine (Itena Obturys) or bioceramic-based sealer (Itena, MTA Bioseal)
Diagnostic Test: PAI Score Comparasion — PAI scores of the patients will be determined with periapical films taken before treatment and compared with oxidative stress markers before and after treatment for the epoxyamine group and bioceramic group.

SUMMARY:
The goal of this clinical trial is to primary purpose investigate and compare oxidative stress markers in patients with chronic apical periodontitis treated with different root canal paste in a single session. The main questions it aims to answer are:

Is there a change in oxidative stress markers measured from saliva after root canal treatment? Is there a difference between the change of oxidative stress markers in patients using different root canal sealers after root canal treatment?

Researchers will compare bioceramic-based and epoxy resin-based root canal sealers to see if there are significant differences in oxidative stress markers measured from patients' saliva after root canal treatment.

* Participants will be informed about all procedures before starting the clinical process.
* Participants are expected to allow saliva sampling two times: first sample will be collected on root canal treatment session and second sample will be collected on the 30th day after root canal treatment.
* Participants will be informed in writing about the treatment procedure before starting the clinical process.
* Participants are expected to sign the informed consent form on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy, ASA1 patients,
* Phase 1 periodontal treatment was performed,
* Diagnosed with chronic apical periodontitis in a single tooth with 2 or more roots in the mouth,
* The lesion measured <2 cm on radiographic evaluation,
* The vitality of the tooth was checked by EPT (Ai-Pex, Woodpecker, China) and Cold test (Cerkamed, Poland) and confirmed to be devitalised,
* Socioculturally able to participate in the treatment,
* Individuals who did not smoke or drink alcohol

Exclusion Criteria:

* Patients who have used antibiotics in the last three months and analgesics in the last two weeks
* Patients who smoke and/or abuse alcohol
* Patients younger than 18 years or older than 45 years,
* Patients with controlled or uncontrolled systemic disease and life-threatening conditions (ASA 2,3,4,5,6)
* Pregnant or lactating women,
* Patients with poor oral hygiene,
* Patients who had head and neck radiotherapy,
* With obesity,
* Active periodontal disease,
* Periodontal pocket depth over 3mm,
* There is enough loss of material in the relevant tooth to prevent adequate isolation or to require post placement,
* Clinical examination of the relevant tooth showing symptoms in percussion-palpation,
* Radiographically, the lesion is seen in relation to anatomical formations such as the mandibular canal and maxillary sinus,
* Patients who required prophylactic antibiotic use before invasive dental procedures were excluded from the study.
* Patients who did not attend the follow-up appointment and patients who experienced complications during expansion (instrument seperation, perforation, etc.) were excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-11-13 (Estimated)

PRIMARY OUTCOMES:
Changes in biochemically measured oxidative stress markers at 30th day in patients treated with epoxyamine/bioceramic root canal pastes. | three month aproximately
  oxidative stress markers (myeloperoxidase, 8-epi, total oxidant status, total antioxidant status, oxidative stress index, malondialdehyde) will be measured and compared biochemically in saliva samples taken from the patients on the first and thirtieth day.
Comparison of the changes observed in biochemically measured oxidative stress markers of patients in the bioceramic group and patients in the epoxyamine group at day 1 and day 30 | three month aproximately
  results of oxidative stress measurement obtained from bioceramic group and epoxyamin group will be compared. comparsion will be performed with biochemical kits for saliva samples.

SECONDARY OUTCOMES:
Investigation of the relationship between biochemically measured oxidative stress markers from endodontium and initial saliva samples obtained from all patients and PAI score determined by periapical films | three months aproximately
  results of PAI and oxidative stress markers measured with biochemical kits will be compromised.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Ordu- Altınordu, Turkey (Türkiye)